CLINICAL TRIAL: NCT00113100
Title: Mechanisms of Skin Repair by Topical Estrogen in Vivo
Brief Title: Mechanisms of Skin Repair by Topical Estrogen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Derm 530
Record Dates: First submitted 2005-06-03; First posted 2005-06-06 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2008-08

CONDITIONS: Skin Wrinkling
Keywords: skin; estrogen; sun damage; Photodamaged Skin
MeSH Terms: interventions — Estradiol; Ethanol; Propylene Glycol

INTERVENTIONS:
Drug: Topical 17-beta estradiol in ethanol/propylene glycol (ETOH/PG)

SUMMARY:
The purpose of this study is to investigate the way by which estrogen improves the appearance of sun damaged human skin. Accumulating evidence suggests that estrogen, taken by post menopausal women, may cause skin to look younger as a consequence of reduced wrinkles. Collagen is the most abundant protein in human skin and gives skin its strength and shape. Recent data indicate that short-term topical estrogen (17-beta estradiol) treatment increases collagen production in sun damaged skin. This study will compare the molecular and microscopic effects from topical 17-beta estradiol (E2) when applied to the skin for a short-term duration. It is anticipated that the new knowledge from this study will enable development of new ways to improve the function of aged skin.

DETAILED DESCRIPTION:
The objectives of the study are to determine if topically-applied 17-beta estradiol (E2), alone or in combination with clobetasol, will produce histological and molecular effects distinguishable from vehicle in human skin. Specifically, the study will focus on regulation of collagen, elastin, and hyaluronic acid production and degradation in human skin, by steroid hormone receptors that are activated by estrogen or clobetasol. The sites to be treated will be buttock, hip, forearm, or facial skin. Subjects will receive between one to twelve vehicle (matching solution without any active ingredients), estrogen, and/or clobetasol topical applications. Skin biopsies of treated areas will be obtained at baseline and at subsequent timepoints. The study will last up to two weeks. Endpoints will include protein and mRNA levels of collagen, elastin, hyaluronic acid, and other components of skin connective tissue. In addition, we will perform cDNA microanalysis to determine estrogen/clobetasol target genes in human skin. The results from our studies will provide new knowledge regarding the molecular basis of skin aging. This new knowledge will enable development of new ways to improve the function of aged skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy post-menopausal (without spontaneous menstrual bleeding for at least 1 year) women, and men, at least 50 years of age and any racial/ethnic type.
* Subjects must understand and sign the informed consent prior to participation.
* Subjects must be in generally good health.
* Subjects must be available for follow-up visits to comply with the requirements of the protocol.
* Not on estrogen replacement therapy within the past 3 months.
* No nonsteroidal anti-inflammatory drugs two weeks prior to study entry.
* No topical steroids two weeks prior to study entry.
* You must live within a reasonable driving distance of Ann Arbor, Michigan, and/or be able to attend all of the scheduled appointments during the study.

Exclusion Criteria:

* History of keloid formation or hypertrophic scarring.
* History of reaction to lidocaine anesthetic.
* Subjects with significant medical history or concurrent condition which the investigator(s) feel is not safe for study participation and which would impair evaluation of test sites.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2004-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Endpoints will include, protein and mRNA levels of collagen, elastin, hyaluronic acid, and other components of skin connective tissue

CONTACTS AND LOCATIONS:
Overall Officials: John J Voorhees, MD, Study Chair — University of Michigan
Locations (1):
- University of Michigan Department of Dermatology, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Rittie L, Kang S, Voorhees JJ, Fisher GJ. Induction of collagen by estradiol: difference between sun-protected and photodamaged human skin in vivo. Arch Dermatol. 2008 Sep;144(9):1129-40. doi: 10.1001/archderm.144.9.1129. PMID 18794456